CLINICAL TRIAL: NCT05728502
Title: A Multi-center, Two-arm, Open-label, Externally Controlled, Post-marketing Study of the Effectiveness and Safety of Vericiguat in HFrEF Patients in China
Brief Title: An Observational Study, Called VERI-China, to Learn More About How Well Vericiguat Works and How Safe it is in Real-world Setting in People With Chronic Heart Failure With Reduced Ejection Fraction (HFrEF) in China
Acronym: VERI-China
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22323
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — vericiguat; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vericiguat arm: Chinese adult patients with Heart Failure with Reduced Ejection Fraction (HFrEF) who are prescribed vericiguat under routine treatment conditions. Data will be prospectively collected.
  Interventions: Drug: Vericiguat (Verquvo, BAY1021189)
- external control arm: Chinese adult HFrEF patients who received SoC treatment will be collected from China Heart Failure Center registry database. This control arm will be retrospectively collected from the patients in the database in the same period, from FPFV to LPFV of the vericiguat arm, and matched by propensity score based on baseline characteristics.
  Interventions: Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: Vericiguat (Verquvo, BAY1021189) — Dosage at the discretion of the treating physician, based on the recommendations written in the product information.
  Groups: vericiguat arm
Drug: Standard of Care (SoC) — Dosage at the discretion of the treating physician.
  Groups: external control arm

SUMMARY:
This is an observational study in which data from people in China with chronic heart failure with reduced ejection fraction (HFrEF) who will be receiving vericiguat treatment are collected. Vericiguat treatment will be compared to available data on standard of care (SOC) treatment. In observational studies, only observations are made without specified advice or interventions.

HFrEF is a long-term condition where the left side of the heart does not pump blood out to the body as well as it should. Blood and fluid may collect in the lungs, blood vessels, and tissues causing shortness of breath or tiredness. Over time, heart failure can lead to other serious medical conditions that may result in hospital stays and death.

The drug vericiguat works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC). The sGC enzyme helps to regulate the heart and blood circulation. Vericiguat is already available in China and other countries for doctors to prescribe to people with heart failure. Vericiguat has already been studied in previous clinical studies. However, the data from these studies were restricted by inclusion and exclusion criteria. Therefore, this real-world study will collect important data from real-world setting in China.

The main purpose of this study is to collect more data on how well vericiguat works compared with current SOC in Chinese people with HFrEF under everyday conditions.

Working well means that the treatment can prevent the following from happening:

* death due to heart and circulatory events,
* a hospital stay due to heart conditions (failure).

In addition, the study team will gather more information about how safe the study drug vericiguat is for Chinese people with HFrEF. To do this, the researchers will collect all medical problems the participants have during the study. These medical problems are also known as "adverse events" and may or may not be related to the study treatment.

Subsequently, the study team will compare the data between participants who received the study drug vericiguat and those who received SOC. The SOC is the currently appropriate treatment in accordance with scientific evidence and agreed upon in collaboration between medical experts for HFrEF.

The participants will take vericiguat as prescribed by their doctors during routine practice according to the approved product information. For the vericiguat group, data will be collected at routine visits, which are not mandated by this study. The data for the comparison (SOC group) will come from a database called China Heart Failure Center. These data will be collected retrospectively for a comparable period of time.

The following data from the study participants will be documented during visits that take place in routine practice every 3 months:

* underlying and concomitant diseases,
* prior medication,
* laboratory parameters,
* vital signs such as blood pressure, heart rate,
* results of cardiac exams (e.g. echocardiography),
* information about how and in which amount vericiguat is usually given to patients.

The participants will be treated with vericiguat and followed up to 12 months or until they leave the study, whatever comes first.

ELIGIBILITY:
Inclusion Criteria:

vericiguat arm

* Female and male patients ≥ 18 years of age who are naïve to vericiguat treatment
* Patients with HFrEF after a recent decompensation episode (within 6 months of heart failure hospitalization or within 3 months of intravenous (IV) diuretics for heart failure not requiring hospitalization)
* Decision to initiate treatment with vericiguat as per the local approved label
* Signed informed consent

control arm

* Aged 18 or over at baseline
* Only patients receiving SoC for chronic heart failure (no history of receiving vericiguat prior to the index date)
* Patients with HFrEF after a recent decompensation episode (within 6 months of heart failure hospitalization or within 3 months of intravenous (IV) diuretics for heart failure not requiring hospitalization)

Exclusion Criteria:

vericiguat arm

* Participation in other investigational program with interventions outside of routine clinical practice
* Contra-indications according to the local marketing authorization label

control arm

* Patients who have started therapy with vericiguat for chronic heart failure at baseline
* Contra-indications according to the vericiguat local marketing authorization label
* Patients participating in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of Chinese adult HFrEF patients who are prescribed vericiguat or standard treatment by the physician.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-12-26 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of the composite of cardiovascular (CV) death or first hospitalization due to Heart Failure (HF) | Up to 1 year.

SECONDARY OUTCOMES:
Time to first occurrence of CV death | Up to 1 year
Time to first occurrence of HF hospitalization | Up to 1 year
Time to first occurrence of the composite of death due to all causes or first HF hospitalization | Up to 1 year
Time to death due to all-causes | Up to 1 year
Occurrence of collected Adverse Event (AE) and Serious Adverse Event (SAE) | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Registries, Multiple Locations, Many Locations, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here for access to information about Bayer's transparency standards and Bayer studies — http://clinicaltrials.bayer.com/